CLINICAL TRIAL: NCT06853977
Title: Understanding the Role of Monoaminergic Neurotransmitters in Cognitive Functions Using Fast-cyclic Voltammetry in Patients With Neurological and Psychiatric Diseases Eligible for Neurosurgical Treatment (COGAMINE)
Acronym: COGAMINE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-A02141-46
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Neurological Diseases or Conditions; Psychiatric Diseases; Candidates for Deep Brain Stimulation; Candidates for Invasive S-EEG; Candidates for Awake Surgery
Keywords: deep brain stimulation; monoaminergic neurotransmitters; awake surgery; Intracerebral FSCV
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intracerebral voltammetric recordings (Experimental)
  Interventions: Behavioral: Cognitive tasks

INTERVENTIONS:
Behavioral: Cognitive tasks — Cognitive tasks performed during intracerebral voltammetric recordings

SUMMARY:
This study aims at dynamically mapping local variations in the concentrations of monoaminergic neurotransmitters (for e.g. dopamine, serotonin and noradrenaline) in the human brain using fast-scan cyclic voltammetric recordings (FSCV). This study will be carried out on patients with neurological (for e.g. brain cancer, Parkinson disease (PD) or treatment-resistant epilepsy …) or psychiatric (for e.g. Treatment resistant obsessive compulsive disorder, depression, Tourette syndrome …) diseases who are eligible to neurosurgical treatment. Typical neurosurgical treatments non-exhaustively include: (1) deep brain stimulation (DBS) electrode implanted as part of the routine management of their pathology (PD, etc.) or as part of clinical trials (treatment resistant depression, resistant obsessive-compulsive disorder, etc.), as well as on patients whose pathology requires invasive exploration by stereotactic-electroencephalography (S-EEG) for therapeutic purposes, either as part of their routine management or as part of a clinical trial. The aim of this mapping is to assess fluctuations in local concentrations of key monoaminergic neurotransmitters involved in cognitive functions at an individual level, with a high temporal (sub-second) and spatial resolution, as well as a sensitivity, that was previously unattainable with other neuroimaging techniques. The data collected in this study will improve our understanding of the role of monoaminergic neurotransmitters in normal human cognition, as well as their dysfunctions in psychiatric and neurological disorders. These data may guide research into new therapeutic targets for the treatment of these pathologies. This study requires a large cohort of patients to build up the most comprehensive database possible, for which access to the information collected is essential.

ELIGIBILITY:
Inclusion Criteria:

* Patient of 18 years old or older;
* Patient undergoing S-EEG invasive exploration OR a neurosurgical procedure (such as DBS or resection neurosurgery in an awake patient) as part of the management of a neurological or psychiatric disease (routine management or participation in a clinical study);
* Patient informed and having signed the consent form;
* Patient able to perform the cognitive tasks proposed.

Exclusion Criteria:

* Patient not affiliated to a social security or other social protection scheme;
* Patient with contraindication to S-EEG or neurosurgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2035-06 (Estimated); Study Completion 2035-06 (Estimated)

PRIMARY OUTCOMES:
Variation in monoaminergic neurotransmitter concentrations | Day 0 to Month 2
  Variation in monoaminergic neurotransmitter concentrations as collected using FSCV during the performance of cognitive tasks in different neuropsychiatric or neuro-oncological pathologies.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalo-Universitaire Paris Psychiatrie & Neurosciences, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mosher CP, Mamelak AN, Malekmohammadi M, Pouratian N, Rutishauser U. Distinct roles of dorsal and ventral subthalamic neurons in action selection and cancellation. Neuron. 2021 Mar 3;109(5):869-881.e6. doi: 10.1016/j.neuron.2020.12.025. Epub 2021 Jan 21. PMID 33482087
- [Background] Hoerl AE, Kennard RW. Ridge Regression: Biased Estimation for Nonorthogonal Problems. Technometrics. 1970;12(1):55-67.
- [Background] Tibshirani R. Regression Shrinkage and Selection Via the Lasso. J R Stat Soc Ser B: Stat Methodol. 2018;58(1):267-88.
- [Background] Zou H, Hastie T. Regularization and Variable Selection Via the Elastic Net. J R Stat Soc Ser B: Stat Methodol. 2005;67(2):301-20.
- [Background] Montague PR, Kishida KT. Computational Underpinnings of Neuromodulation in Humans. Cold Spring Harb Symp Quant Biol. 2018;83:71-82. doi: 10.1101/sqb.2018.83.038166. Epub 2019 Apr 25. PMID 31023828
- [Background] Gogos AJ, Young JS, Morshed RA, Hervey-Jumper SL, Berger MS. Awake glioma surgery: technical evolution and nuances. J Neurooncol. 2020 May;147(3):515-524. doi: 10.1007/s11060-020-03482-z. Epub 2020 Apr 8. PMID 32270374
- [Background] Matthews J, Nagao K, Ding C, Newby R, Kempster P, Hohwy J. Raised visual contrast thresholds with intact attention and metacognition in functional motor disorder. Cortex. 2020 Apr;125:161-174. doi: 10.1016/j.cortex.2019.12.009. Epub 2020 Jan 3. PMID 31991241
- [Background] Huang YT, Georgiev D, Foltynie T, Limousin P, Speekenbrink M, Jahanshahi M. Different effects of dopaminergic medication on perceptual decision-making in Parkinson's disease as a function of task difficulty and speed-accuracy instructions. Neuropsychologia. 2015 Aug;75:577-87. doi: 10.1016/j.neuropsychologia.2015.07.012. Epub 2015 Jul 13. PMID 26184442
- [Background] Volkow ND, Fowler JS, Gatley SJ, Logan J, Wang GJ, Ding YS, Dewey S. PET evaluation of the dopamine system of the human brain. J Nucl Med. 1996 Jul;37(7):1242-56. PMID 8965206
- [Background] Ng J, Papandreou A, Heales SJ, Kurian MA. Monoamine neurotransmitter disorders--clinical advances and future perspectives. Nat Rev Neurol. 2015 Oct;11(10):567-84. doi: 10.1038/nrneurol.2015.172. Epub 2015 Sep 22. PMID 26392380
- [Background] Bergman H. The Hidden Life of the Basal Ganglia: At the Base of Brain and Mind. 2021.
- [Background] Tye KM, Deisseroth K. Optogenetic investigation of neural circuits underlying brain disease in animal models. Nat Rev Neurosci. 2012 Mar 20;13(4):251-66. doi: 10.1038/nrn3171. PMID 22430017
- [Background] Bucher ES, Wightman RM. Electrochemical Analysis of Neurotransmitters. Annu Rev Anal Chem (Palo Alto Calif). 2015;8:239-61. doi: 10.1146/annurev-anchem-071114-040426. Epub 2015 May 4. PMID 25939038
- [Background] Nutt DJ, Lingford-Hughes A, Erritzoe D, Stokes PR. The dopamine theory of addiction: 40 years of highs and lows. Nat Rev Neurosci. 2015 May;16(5):305-12. doi: 10.1038/nrn3939. Epub 2015 Apr 15. PMID 25873042
- [Background] Otte C, Gold SM, Penninx BW, Pariante CM, Etkin A, Fava M, Mohr DC, Schatzberg AF. Major depressive disorder. Nat Rev Dis Primers. 2016 Sep 15;2:16065. doi: 10.1038/nrdp.2016.65. PMID 27629598
- [Background] Craske MG, Stein MB, Eley TC, Milad MR, Holmes A, Rapee RM, Wittchen HU. Anxiety disorders. Nat Rev Dis Primers. 2017 May 4;3:17024. doi: 10.1038/nrdp.2017.24. PMID 28470168
- [Background] Dayan P. Twenty-five lessons from computational neuromodulation. Neuron. 2012 Oct 4;76(1):240-56. doi: 10.1016/j.neuron.2012.09.027. PMID 23040818
- [Background] Boureau YL, Dayan P. Opponency revisited: competition and cooperation between dopamine and serotonin. Neuropsychopharmacology. 2011 Jan;36(1):74-97. doi: 10.1038/npp.2010.151. Epub 2010 Sep 29. PMID 20881948
- [Background] Marder E. Neuromodulation of neuronal circuits: back to the future. Neuron. 2012 Oct 4;76(1):1-11. doi: 10.1016/j.neuron.2012.09.010. PMID 23040802
- [Background] Kandel ER, Koester JD, Mack SH, Siegelbaum SA. Principles of neural science, 6th ed. Hill MG, editor. 2021.
- [Background] Portas CM, Bjorvatn B, Ursin R. Serotonin and the sleep/wake cycle: special emphasis on microdialysis studies. Prog Neurobiol. 2000 Jan;60(1):13-35. doi: 10.1016/s0301-0082(98)00097-5. PMID 10622375
- [Background] Must A, Juhasz A, Rimanoczy A, Szabo Z, Keri S, Janka Z. Major depressive disorder, serotonin transporter, and personality traits: why patients use suboptimal decision-making strategies? J Affect Disord. 2007 Nov;103(1-3):273-6. doi: 10.1016/j.jad.2007.02.001. Epub 2007 Mar 26. PMID 17382402
- [Background] Diekhof EK, Falkai P, Gruber O. Functional neuroimaging of reward processing and decision-making: a review of aberrant motivational and affective processing in addiction and mood disorders. Brain Res Rev. 2008 Nov;59(1):164-84. doi: 10.1016/j.brainresrev.2008.07.004. Epub 2008 Jul 21. PMID 18675846
- [Background] Yildiz O, Smith JR, Purdy RE. Serotonin and vasoconstrictor synergism. Life Sci. 1998;62(19):1723-32. doi: 10.1016/s0024-3205(97)01166-1. PMID 9585103
- [Background] Goldstein DS. Catecholamines in the periphery. Overview. Adv Pharmacol. 1998;42:529-39. doi: 10.1016/s1054-3589(08)60806-6. No abstract available. PMID 9327957
- [Background] Moran RJ, Kishida KT, Lohrenz T, Saez I, Laxton AW, Witcher MR, Tatter SB, Ellis TL, Phillips PE, Dayan P, Montague PR. The Protective Action Encoding of Serotonin Transients in the Human Brain. Neuropsychopharmacology. 2018 May;43(6):1425-1435. doi: 10.1038/npp.2017.304. Epub 2018 Jan 3. PMID 29297512
- [Background] Sands LP, Jiang A, Liebenow B, DiMarco E, Laxton AW, Tatter SB, Montague PR, Kishida KT. Subsecond fluctuations in extracellular dopamine encode reward and punishment prediction errors in humans. Sci Adv. 2023 Dec;9(48):eadi4927. doi: 10.1126/sciadv.adi4927. Epub 2023 Dec 1. PMID 38039368
- [Background] Kishida KT, Saez I, Lohrenz T, Witcher MR, Laxton AW, Tatter SB, White JP, Ellis TL, Phillips PE, Montague PR. Subsecond dopamine fluctuations in human striatum encode superposed error signals about actual and counterfactual reward. Proc Natl Acad Sci U S A. 2016 Jan 5;113(1):200-5. doi: 10.1073/pnas.1513619112. Epub 2015 Nov 23. PMID 26598677
- [Background] Kishida KT, Sandberg SG, Lohrenz T, Comair YG, Saez I, Phillips PE, Montague PR. Sub-second dopamine detection in human striatum. PLoS One. 2011;6(8):e23291. doi: 10.1371/journal.pone.0023291. Epub 2011 Aug 4. PMID 21829726
- [Background] Bang D, Kishida KT, Lohrenz T, White JP, Laxton AW, Tatter SB, Fleming SM, Montague PR. Sub-second Dopamine and Serotonin Signaling in Human Striatum during Perceptual Decision-Making. Neuron. 2020 Dec 9;108(5):999-1010.e6. doi: 10.1016/j.neuron.2020.09.015. Epub 2020 Oct 12. PMID 33049201
- [Background] Liebenow B, Jiang A, DiMarco E, Wilson T, Siddiqui MS, Ul Haq I, Laxton AW, Tatter SB, Kishida KT. Intracranial subsecond dopamine measurements during a "sure bet or gamble" decision-making task in patients with alcohol use disorder suggest diminished dopaminergic signals about relief. Neurosurg Focus. 2023 Feb;54(2):E3. doi: 10.3171/2022.11.FOCUS22614. PMID 36724520
- [Background] Clark JJ, Sandberg SG, Wanat MJ, Gan JO, Horne EA, Hart AS, Akers CA, Parker JG, Willuhn I, Martinez V, Evans SB, Stella N, Phillips PE. Chronic microsensors for longitudinal, subsecond dopamine detection in behaving animals. Nat Methods. 2010 Feb;7(2):126-9. doi: 10.1038/nmeth.1412. Epub 2009 Dec 27. PMID 20037591